CLINICAL TRIAL: NCT05310435
Title: A New Intelligent Stocking for Quantification of Edema in the Lower Limbs
Status: Terminated | Type: Observational
Why Stopped: Not enough patients
Sponsor: University of Aarhus (Other)
Collaborators: Ohmatex ApS (Unknown); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Alexander Emil Kaspersen, Project manager, University of Aarhus
Other Study IDs: 1-10-72-143-17; 2017084027 (Other: Danish Medicines Agency)
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Edema Leg
Keywords: Lower leg edema; Equivalence study; Leg volume

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women with lower leg edema: Pregnant women with clinical lower leg edema measured two times with Edema Stocking device, two times with water displacement volumetry and two with tape measure each day for three days.
  Interventions: Device: Single volume measurement with ESD; Device: Single volume measurement with WDV; Device: Single circumference measurement with tape measure; Device: Continuous volume measurement with ESD

INTERVENTIONS:
Device: Single volume measurement with ESD — Single volume measurement with Edema Stocking device
Device: Single volume measurement with WDV — Single volume measurement with water displacement volumetry method
Device: Single circumference measurement with tape measure — Single circumference measurement with tape measure
Device: Continuous volume measurement with ESD — Continuous volume measurement with Edema Stocking device

SUMMARY:
The purpose of the study is to evaluate a prototype of an intelligent stocking (Edema Stocking Device [ESD]), consisting of two stretch sensitive sensors, as a new method for continuously lower leg volume monitoring. The study is a scientific evaluation of the ESD compared with water displacement volumetry and tape measure.

DETAILED DESCRIPTION:
Background:

Balance of body fluids is strictly regulated within a narrow range and is controlled by water movement between the interstitial compartment and the capillaries. An unnatural balance between the two compartments can be seen in several diseases, leading to a net filtration out of the vascular space, resulting in the formation of edema. Monitoring of edema formation represents a unique way of evaluating the degree of the underlying disease and effect of treatment. Numerous different methods can be used to quantify leg volume. However, no current method provides continuous quantitative assessment. The feasibility of continuous lower leg measuring using an intelligent stocking was hypothesized.

The aim of the study was to evaluate the Edema Stocking device (ESD) as a tool for continuous quantification of edema compared with water displacement volumetry (WDV) and tape measure.

Materials and methods:

Study design: Non-randomized equivalence study. Experimental comparison study of new method compared to golden standard.

ELIGIBILITY:
Inclusion Criteria:

* Edema of the lower legs.
* Between 20-18 years.
* Identified at Department of Gynaecology and Obstetrics, Aarhus University Hospital, Denmark.

Exclusion Criteria:

* Length of lower leg of more than 34,0 cm (measured from floor to knee).

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women, 20-40 years, located to the Central Region of Denmark, admitted to Department of Gynaecology and Obstetrics, Aarhus University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Leg volume measured with ESD (ml) | 1 minute
  Obtained with the Edema Stocking device
Leg volume measured with WDV (ml) | 1 minute
  Obtained with water displacement volumetry
Leg circumference measured with tape measure (mm) | 1 minute
  Obtained with tape measure
Leg circumference measured with ESD (mm) | 60 minutes
  Obtained with the Edema Stocking Device

CONTACTS AND LOCATIONS:
Overall Officials: Olav B Petersen, MD, PhD, Study Director — Aarhus University Hospital
Locations (1):
- Department og Gynaecology and Obstetrics, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT05310435/ICF_000.pdf